CLINICAL TRIAL: NCT03250000
Title: Changes in Microcirculation and Functional Status During Exacerbation of COPD
Acronym: COPD-EX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Martijn Spruit, PhD, Hasselt University
Other Study IDs: COPD-EX HasseltU
Record Dates: First submitted 2017-06-21; First posted 2017-08-15 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: COPD Exacerbation; Physical Activity; Retinal Vascular
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD-stable: Stable COPD patients at pulmonology consultation in Ziekenhuis Oost-Limburg (ZOL) Genk
- COPD-Ex: Patients admitted to the respiratory ward of ZOL Genk with a diagnosis of acute exacerbation, based on the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria.

SUMMARY:
This study investigates the influence of acute exacerbation of chronic obstructive pulmonary disease (COPD) on retinal microcirculation, on functional status and also investigates the prognostic value of retinal vessel caliber assessment in terms of hospitalization and mortality during 2 years of follow-up.

DETAILED DESCRIPTION:
Recent findings suggest that patients with chronic obstructive pulmonary disease (COPD) are at increased risk for myocardial infarction and stroke during periods of acute exacerbation. These findings might be related to acute endothelial changes associated to increased systemic inflammation. Changes in the microcirculation can be explored noninvasively by studying retinal blood vessels that are visualized in fundus images. The retinal blood vessels have anatomical and physiological features that are comparable with the coronary circulation.

Patients with COPD experience quadriceps muscle weakness, which worsens during hospitalization by ~1% per day. This is the result of physical inactivity, in combination with increased oxidative stress and systemic inflammation. Physical inactivity is induced by the hospital environment, but is also related to symptoms of dyspnea caused by increased work of breathing and oxygen desaturation.

Muscle weakness and physical inactivity are associated to poor functional status and recurrent hospital admissions, independent of pulmonary impairment, which makes those patients with frequent exacerbations prone to enter a vicious cycle.

Simple functional screening tests during hospital stay might enable us to quantify the impact of a hospitalization on functional status and to identify patients at risk for repeated exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD (post-bronchodilator forced expiratory volume / forced vital capacity < 0.7), no exacerbations in the previous weeks. COPD patients with diagnosis of acute exacerbation, based on the GOLD criteria.

Exclusion Criteria:

* Inability to walk without support from others

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable and exacerbated COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Retinal microcirculation | Stable: Outpatient clinic/ COPD exacerbated: Day 2-3 in hospital; Day 5-7 in hospital; 4 weeks after discharge
  Fundus of the right eye will be photographed using a retinal camera. The vessel diameters had geometric patterns will be measure.
Changes in Functional status tests | Stable: Outpatient clinic/ COPD exacerbated: Day 2-3 in hospital; Day 5-7 in hospital; 4 weeks after discharge
  Short physical performance battery (SPPB), which consists of a four meter gait test, a five-repetition sit-to-stand test and a balance test will be done. All the testes ranged from 0 to 4 and the sum of the three components comprised the final SPPB score, with a possible range from 0 to 12.

SECONDARY OUTCOMES:
Functional exercise tolerance | Stable: Outpatient clinic/ COPD exacerbated: Day 2-3 in hospital; Day 5-7 in hospital; 4 weeks after discharge
  Six minute walk test will be done
Muscle Function | Stable: Outpatient clinic/ COPD exacerbated: Day 2-3 in hospital; Day 5-7 in hospital; 4 weeks after discharge
  Handgrip and Isometric-eccentric quadriceps strength test will be done
Changes in Daily physical activity | Stable: Outpatient clinic/ COPD exacerbated: Day 2-3 in hospital; Day 5-7 in hospital; 4 weeks after discharge
  Activity level will be assess by an accelerometer, the patient will be worn for 7 days.
Impact of the disease | Stable: Outpatient clinic/ COPD exacerbated: Day 2-3 in hospital; Day 5-7 in hospital; 4 weeks after discharge
  The COPD assessment test will be applied
Impact of the dyspnea | Stable: Outpatient clinic/ COPD exacerbated: Day 2-3 in hospital; Day 5-7 in hospital; 4 weeks after discharge
  The modified medical research council scale will be applied
Impact of the depression | Stable: Outpatient clinic/ COPD exacerbated: Day 2-3 in hospital; Day 5-7 in hospital; 4 weeks after discharge
  The patient health questionnaire will be applied
Impact of the fatigue | Stable: Outpatient clinic/ COPD exacerbated: Day 2-3 in hospital; Day 5-7 in hospital; 4 weeks after discharge
  The checklist individual strength- fatigue sub-scale will be applied
Body composition | Stable: Outpatient clinic/ COPD exacerbated: Day 2-3 in hospital; Day 5-7 in hospital; 4 weeks after discharge
  Bio-electrical impedance analysis will be used to estimate fat-free body mass based on the assessment of total body water. Body mass index and waist circumference will provide general information about body composition.
Cardiovascular parameters | Stable: Outpatient clinic/ COPD exacerbated: Day 2-3 in hospital; Day 5-7 in hospital; 4 weeks after discharge
  Resting ankle and brachial blood pressure will be measured and the ankle brachial pressure index will be calculated by the ratio of ankle to ipsilateral brachial systolic blood pressure
Continuous assessment of oxygen saturation | COPD exacerbated: Day 5-7 in hospital; 4 weeks after discharge
  A portable pulse oximeter will be worn to asses transcutaneous oxygen saturation for 24 hours in patients with an exacerbation.
Continuous assessment of heart rate | COPD exacerbated: Day 5-7 in hospital; 4 weeks after discharge
  A portable pulse oximeter will be worn to asses heart rate for 24 hours in patients with an exacerbation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No